CLINICAL TRIAL: NCT04771468
Title: "Hemodynamic Changes During Endovascular Revascularization for Acute Stroke. An Observational Study".
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Collaborators: Ospedale Policlinico San Martino (Other)
Responsible Party: Sponsor
Other Study IDs: STROKE_EMO
Record Dates: First submitted 2021-01-06; First posted 2021-02-25 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sovratentorial ischemic stroke
  Interventions: Device: MOSTCAREup Monitoring; Device: Ecocardiography

INTERVENTIONS:
Device: MOSTCAREup Monitoring — The patients will be equipped with mini-invasive hemodynamic monitoring (the MOSTACAREup system). The MOSTCAREup obtains the hemodynamic data from either the same arterial femoral line used by the neuro-radiologist to perform the treatment or from a dedicated radial artery, as decided by the attending anesthetist to monitor and optimize arterial pressure (the decision to use the arterial line is at discretion of the attending anesthetist for clinical reasons and does not delay the procedure, which starts using always the femoral access).
Device: Ecocardiography — Echocardiography will be performed 1) soon after the end of the treatment (whenever possible, avoiding delays, before od during the treatment in the angiography room); 2) at day 1 after the procedure; 3) at day 3 after the procedure.

SUMMARY:
Neurocardiology is an emerging specialty that addresses the interaction between the brain and the heart, i.e. the effects of cardiac injury on the brain, and the effects of brain injury on the heart. Accumulating clinical and experimental evidence suggests a causal relationship between brain damage and heart dysfunction.

ELIGIBILITY:
Inclusion criteria

1. Adult patients aged ≥ 18 years.
2. Acute supratentorial or carotid stroke. Exclusion criteria

1. Invasive arterial signal unsuitable to obtain hemodynamic data. 2. Emergency neurosurgery needed before intra-arterial treatment. 3. Once enrolled, the patient can be excluded from the study because of one of the following intraoperative conditions:

1. Intraoperative technical limitations limiting or impeding the arterial re-opening
2. Persistent low quality of the arterial signal. After positioning the patient and zeroing the arterial signal, the arterial waveform is checked for quality by means of a square-wave test and optimized in the case of the occurrence of under or over-damping.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted for acute ischemic stroke
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac output measurement | Up to 6 hours after clot removal
  Changes of cardiac output of the enrolled patients before and after clot removal.
Arterial elastance measurement | Up to 6 hours after clot removal
  Changes of arterial elastance of the enrolled patients before and after clot removal.
Arterial blood pressure measurement | Up to 6 hours after clot removal
  Changes of arterial blood pressure of the enrolled patients before and after clot removal.
Heart rate variability measurement | Up to 6 hours after clot removal
  Changes of heart rate variability of the enrolled patients before and after clot removal.

SECONDARY OUTCOMES:
Transthoracic echocardiography | at the admission
  Ejection Fraction measurement
Transthoracic Echocardiography | up to 3 weeks after clot removal
  wave E assessment
Transthoracic Echocardiography | up to 3 weeks after clot removal
  wave A assessment
Transthoracic Echocardiography | up to 3 weeks after clot removal
  wave e' assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study will be available from the corresponding author on reasonable request.